CLINICAL TRIAL: NCT02584062
Title: The Eye Hospital of Tianjin Medical University
Brief Title: Clinical Observation of Technologic Application of No-touch Fluid-air Exchange in Surgery of Idiopathic Macula Hole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Bojie Hu, Head of Ophthalmology department, Principal Investigator, Associate Senior Physician, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBJ 151617
Record Dates: First submitted 2015-10-09; First posted 2015-10-22 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Idiopathic Macula Hole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- no-touch fluid-air exchange group (Experimental): All patients in no-touch fluid-air exchange group will have a surgery of vitrectomy metrectomy and internal membrane peeling and gas tamponed.In this surgery ,investigator will not touch the macular area,especially the area of the macular hole and investigator will not have the fluid-air exchange of the macular area.
  Interventions: Procedure: no-touch fluid-air exchange; Procedure: vitrectomy metrectomy and internal membrane peeling and gas tamponed
- the tradional group (Experimental): All patients in no-touch fluid-air exchange group will have a surgery of vitrectomy metrectomy and internal membrane peeling and gas tamponed.In this surgery ,investigator will touch the macular area and investigator will have the fluid-air exchange.
  Interventions: Procedure: vitrectomy metrectomy and internal membrane peeling and gas tamponed

INTERVENTIONS:
Procedure: no-touch fluid-air exchange
  Other Names: vitrectomy metrectomy and internal membrane peeling and gas tamponed
  Arms: no-touch fluid-air exchange group
Procedure: vitrectomy metrectomy and internal membrane peeling and gas tamponed

SUMMARY:
The purpose of this study is to observe the technologic application of no-touch fluid-air exchange in Surgery of Idiopathic Macula Hole.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed as having an idiopathic macular hole(IMH) by Optical Coherence Tomography(OCT).

Exclusion Criteria:

* Myopia of >6 diopters
* Ocular trauma and other systematic or ocular issues associated with IMHs，such as the other macula disease, for example the degeneration of macula.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
the closure rate of Macular hole | one month
  the closure rate of macular hole through OCT
the closure rate of Macular hole | three month
  the closure rate of Macular hole
the closure rate of Macular hole | six month
  the closure rate of Macular hole

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China